CLINICAL TRIAL: NCT01782495
Title: Open-Label, Phase 2 Study to Evaluate the Safety and Efficacy of the Combination of ABT-450/Ritonavir/ABT-267 With ABT-333 and With or Without RBV in HCV Genotype 1 and ABT-450/r/ABT-267 With RBV in HCV GT4-Infected Adult Liver or Renal Transplant Recipients With Hepatitis C Virus (HCV) Infection (CORAL-I)
Brief Title: A Study to Evaluate Chronic Hepatitis C Infection in Adult Transplant Recipients
Acronym: CORAL-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-999; 2012-004792-39 (EudraCT Number)
Record Dates: First submitted 2013-01-22; First posted 2013-02-04 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C Genotype 4; Chronic Hepatitis; Interferon-Free; Hepatitis C Virus (HCV); Renal Transplant; Liver Transplant; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Arm A (Experimental): Liver transplant recipients with HCV genotype 1 infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm B (Experimental): Liver transplant recipients with HCV genotype 1a or genotype 1b (dependent on prior treatment experience and response) infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm C (Experimental): Liver transplant receipts with HCV genotype 1b infection who were treatment naïve or prior responders to interferon treatment without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) for 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir
- Arm D (Experimental): Liver transplant recipients with HCV genotype 1a infection with Child Pugh A cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (dosed 1,000 or 1,200 mg daily divided twice a day) for 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm E (Experimental): Liver transplant recipients with HCV genotype 1b infection with Child Pugh A cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm F (Experimental): Liver transplant recipients with HCV genotype 1a infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm G (Experimental): Liver transplant recipients with HCV genotype 1b infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir
- Arm H (Experimental): Renal transplant recipients with HCV genotype 1a infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin
- Arm I (Experimental): Renal transplant recipients with HCV genotype 1b infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir
- Arm J (Experimental): Liver transplant recipients with HCV genotype 4 infection without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin
- Arm K (Experimental): Liver transplant recipients with HCV genotype 4 infection with Child Pugh A cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) plus weight-based ribavirin (1,000 or 1,200 mg daily divided twice a day) for 24 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
  Arms: Arm A; Arm B; Arm C; Arm D; Arm E; Arm F; Arm G; Arm H; Arm I
Drug: ombitasvir/paritaprevir/ritonavir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir
  Other Names: TECHNIVIE; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267
  Arms: Arm J; Arm K
Drug: ribavirin — tablet
  Arms: Arm A; Arm B; Arm D; Arm E; Arm F; Arm H; Arm J; Arm K

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-450/r/ABT-267 with or without ABT-333 and with or without ribavirin (RBV) in adult liver or renal transplant recipients with hepatitis C virus (HCV) genotype 1 or 4 (GT1 or GT4) infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at the time of screening.
* Currently taking an immunosuppressant regimen based on either tacrolimus or cyclosporine. Corticosteroids such as prednisone or prednisolone are permitted as components of the immunosuppressant regimen providing the dose is not more than 10 mg/day.
* Hepatitis C virus (HCV) interferon (IFN) therapy treatment-naïve or -experienced, either pre- or post-liver or renal transplant.
* Screening HCV genotype testing indicating infection with genotype 1 or 4 (GT1 or GT4) only.

Exclusion Criteria:

* Use of everolimus or sirolimus as part of the immunosuppressive regimen within 2 months of Screening Visit.
* Use of any medications contraindicated for use with the study regimen as well as those that are contraindicated for use with either ritonavir or ribavirin within 2 weeks prior to study drugs administration or 10 half-lives (if known), whichever is longer.
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* Documented history of post-transplant complications directly involving the hepatic or renal vasculature as appropriate to the organ transplanted, e.g., thrombosis of the portal vein, the hepatic artery and/or hepatic vein.
* Clinically significant abnormalities, other than HCV infection, in a subject post-transplant based upon the medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG) that make the subject an unsuitable candidate for this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Kwo PY, Mantry PS, Coakley E, Te HS, Vargas HE, Brown R Jr, Gordon F, Levitsky J, Terrault NA, Burton JR Jr, Xie W, Setze C, Badri P, Pilot-Matias T, Vilchez RA, Forns X. An interferon-free antiviral regimen for HCV after liver transplantation. N Engl J Med. 2014 Dec 18;371(25):2375-82. doi: 10.1056/NEJMoa1408921. Epub 2014 Nov 11. PMID 25386767
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 35-day screening period.
Groups:
- Arm C: Liver transplant receipts with HCV 1b infection who were treatment naïve or prior responders to interferon treatment without cirrhosis received ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) for 24 weeks.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Started | 34 | 27 | 13 | 4 | 2 | 22 | 12 | 9 | 3 | 2 | 1
Completed | 34 | 26 | 13 | 4 | 2 | 22 | 12 | 6 | 3 | 2 | 1
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K | Total
Number analyzed (Participants) | 34 | 27 | 13 | 4 | 2 | 22 | 12 | 9 | 3 | 2 | 1 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (6.62) | 58.0 (6.66) | 61.8 (5.76) | 59.8 (10.78) | 78.0 (1.41) | 58.3 (9.35) | 62.2 (7.64) | 58.0 (8.00) | 57.3 (9.29) | 63.5 (7.78) | 50.0 (NA) — The estimated standard deviation of one sample is undefined | 59.6 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 5 | 0 | 2 | 2 | 2 | 2 | 1 | 0 | 0 | 25
  Male | 27 | 23 | 8 | 4 | 0 | 20 | 10 | 7 | 2 | 2 | 1 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. Participants with missing data after backward imputation were imputed as nonresponders.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 34 | 27 | 13 | 4 | 2 | 22 | 12 | 9 | 3 | 2 | 1
percentage of participants | 97.1 [85.1 to 99.5] | 96.3 [81.7 to 99.3] | 100 [77.2 to 100.0] | 100 [51.0 to 100.0] | 100 [34.2 to 100.0] | 95.5 [78.2 to 99.2] | 100 [75.8 to 100.0] | 66.7 [35.4 to 87.9] | 100 [43.9 to 100.0] | 100 [34.2 to 100.0] | 100 [20.7 to 100.0]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-treatment (SVR24)
Description: SVR24 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 24 weeks after the last dose of study drug. Participants with missing data after backward imputation were imputed as nonresponders.
Time Frame: 24 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 34 | 27 | 13 | 4 | 2 | 22 | 12 | 9 | 3 | 2 | 1
percentage of participants | 97.1 [85.1 to 99.5] | 96.3 [81.7 to 99.3] | 100 [77.2 to 100.0] | 100 [51.0 to 100.0] | 100 [34.2 to 100.0] | 95.5 [78.2 to 99.2] | 100 [75.8 to 100.0] | 66.7 [35.4 to 87.9] | 100 [43.9 to 100.0] | 100 [34.2 to 100.0] | 100 [20.7 to 100.0]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment, or confirmed HCV RNA ≥ LLOQ at any point during treatment after HCV RNA < LLOQ, or HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks (≥ 36 days) of treatment.
Time Frame: Up to 12 weeks (for 12-week treatment) or 24 weeks (for 24-week treatment)
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 34 | 27 | 13 | 4 | 2 | 22 | 12 | 9 | 3 | 2 | 1
percentage of participants | 0 [0.0 to 10.2] | 3.7 [0.7 to 18.3] | 0 [0.0 to 22.8] | 0 [0.0 to 49.0] | 0 [0.0 to 65.8] | 0 [0.0 to 14.9] | 0 [0.0 to 24.2] | 0 [0.0 to 29.9] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 79.3]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 33 | 26 | 12 | 4 | 2 | 21 | 12 | 6 | 3 | 2 | 1
percentage of participants | 3.0 [0.5 to 15.3] | 0 [0.0 to 12.9] | 0 [0.0 to 24.2] | 0 [0.0 to 49.0] | 0 [0.0 to 65.8] | 4.8 [0.8 to 22.7] | 0 [0.0 to 24.2] | 0 [0.0 to 39.0] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 79.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 30 days after the last dose of study drug. TEAEs and TESAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E | ARM F | ARM G | ARM H | ARM I | ARM J | ARM K
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/27 | 0/13 | 0/4 | 0/2 | 0/22 | 0/12 | 1/9 | 0/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/34 | 1/27 | 0/13 | 0/4 | 0/2 | 2/22 | 1/12 | 4/9 | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 33/34 | 27/27 | 12/13 | 4/4 | 2/2 | 22/22 | 12/12 | 8/9 | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=34) | ARM B (N=27) | ARM C (N=13) | ARM D (N=4) | ARM E (N=2) | ARM F (N=22) | ARM G (N=12) | ARM H (N=9) | ARM I (N=3) | ARM J (N=2) | ARM K (N=1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=34) | ARM B (N=27) | ARM C (N=13) | ARM D (N=4) | ARM E (N=2) | ARM F (N=22) | ARM G (N=12) | ARM H (N=9) | ARM I (N=3) | ARM J (N=2) | ARM K (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 8 | 8 | 1 | 3 | 2 | 4 | 0 | 2 | 1 | 0 | 0
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EYE PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OCULAR DISCOMFORT (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OCULAR HYPERAEMIA (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VITREOUS FLOATERS (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANAL PRURITUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BOWEL MOVEMENT IRREGULARITY (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 1
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 9 | 6 | 1 | 1 | 1 | 6 | 2 | 2 | 0 | 0 | 0
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 8 | 11 | 2 | 2 | 1 | 4 | 0 | 2 | 0 | 0 | 0
OESOPHAGEAL DILATATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TOOTH IMPACTED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 4 | 5 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
ASTHENIA (General disorders) | 8 | 7 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHILLS (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EXERCISE TOLERANCE DECREASED (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FACE OEDEMA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 17 | 14 | 4 | 4 | 0 | 14 | 2 | 6 | 1 | 1 | 1
FEELING ABNORMAL (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FEELING COLD (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERNIA PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 5 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
PAIN (General disorders) | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LIVER TRANSPLANT REJECTION (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FUNGAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HORDEOLUM (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINEA CRURIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
POST-TRAUMATIC NECK SYNDROME (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SCRATCH (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUNBURN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUPERFICIAL INJURY OF EYE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD URINE PRESENT (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CARDIAC MURMUR (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATOCRIT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
IMMUNOSUPPRESSANT DRUG LEVEL INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VITAMIN D DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
WEIGHT DECREASED (Investigations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WEIGHT INCREASED (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 3 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE FATIGUE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 6 | 4 | 1 | 1 | 1 | 4 | 2 | 1 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 15 | 8 | 2 | 2 | 1 | 6 | 6 | 3 | 0 | 0 | 0
HYPERSOMNIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
POOR QUALITY SLEEP (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SEIZURE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUNNEL VISION (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AFFECT LABILITY (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APATHY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EMOTIONAL DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 9 | 3 | 0 | 1 | 1 | 3 | 2 | 2 | 0 | 0 | 0
IRRITABILITY (Psychiatric disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
LIBIDO INCREASED (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NIGHTMARE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
POLYURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GENITAL RASH (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PENILE BLISTER (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHOKING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 2 | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 0
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 4 | 2 | 5 | 4 | 1 | 0 | 1 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 7 | 9 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SKIN TIGHTNESS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.